CLINICAL TRIAL: NCT00267800
Title: Registration of Clinical Data and DNA/Serum of Patients With Interstitial Lung Diseases (ILD)
Brief Title: Database of Interstitial Lung Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St. Antonius Hospital (Other)
Other Study IDs: R05.08/A
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2005-12

CONDITIONS: Interstitial Lung Diseases
Keywords: Lung disease, Interstitial; Sarcoidosis; Pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Sarcoidosis; Pulmonary Fibrosis

SUMMARY:
The cause of most interstitial lung diseases (ILDs) is still unknown. Further research, for example to determine predisposing genetic factors, is therefore needed. A database with relevant clinical data and DNA/serum samples of ILD patients could facilitate future research on the cause of ILDs.

DETAILED DESCRIPTION:
Protocol title: 'Registration of clinical data and DNA of patients with Interstitial Lung Disease (ILD)' Rationale: The etiopathogenesis of most Interstitial Lung Diseases (ILDs) is still unknown. Further research, e.g. to determine predisposing genetic factors, is therefore needed. A database with relevant clinical data and DNA/serum samples of ILD patients could facilitate future research on the etiopathogenesis of ILDs.

Objective: Availability of relevant clinical data and DNA/serum samples of ILD patients in a database. Those data can be used for future research.

Study design: A prospective observational study

Study population: Patients diagnosed with ILD attending the pulmonology department in participating hospitals.

Intervention: a blood sample is taken from each patient. Furthermore, additional information is collected from the medical file.

Main study parameters/endpoints: DNA and serum sample, demographic variables, medical information, occupational history and hobbies.

Nature and extent of the burden and risks associated with participation, group relatedness: two tubes of blood will be drawn from the patients. The risks of drawing blood from a vein are minimal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an ILD, as stated by the American Thoracic Society (ATS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100000
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: J.M.M. van den Bosch, M.D., Principal Investigator — St. Antonius Hospital; J.C. Grutters, M.D., Principal Investigator — St. Antonius Hospital
Locations (4):
- Netherlands (4):
  - St. Antonius Hospital, Nieuwegein
  - Diakonessenhuis, Utrecht
  - Mesos Medisch Centrum, Utrecht
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Drent M, Wijnen PA, Jessurun NT, Harmsze AM, Bekers O, Bast A. Drug-Gene Risk Stratification in Patients with Suspected Drug-Induced Interstitial Lung Disease. Drug Saf. 2024 Apr;47(4):355-363. doi: 10.1007/s40264-024-01400-0. Epub 2024 Mar 9. PMID 38460070
- [Derived] Jessurun NT, Drent M, Wijnen PA, Harmsze AM, van Puijenbroek EP, Bekers O, Bast A. Role of Drug-Gene Interactions and Pharmacogenetics in Simvastatin-Associated Pulmonary Toxicity. Drug Saf. 2021 Nov;44(11):1179-1191. doi: 10.1007/s40264-021-01105-8. Epub 2021 Oct 4. PMID 34606062